CLINICAL TRIAL: NCT02829424
Title: Multicenter Randomized Double Blind Controlled-study to Assess the Potential of Methotrexate Versus Placebo to Improve and Maintain Response to Anti TNF- Alpha Agents in Adult Patients With Moderate to Severe Psoriasis
Acronym: METHOBIO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: new treatment on the market in direct competition with the new treatment proposed by the study. Recruitment difficulties.
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-50; 2015-003891-54 (EudraCT Number)
Record Dates: First submitted 2016-06-30; First posted 2016-07-12 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Use of low dose methotrexate (MTX) in psoriasis patients receiving an anti TNF alpha agent according to the approved indication: etanercept- Enbrel®, adalimumab- Humira ®, infliximab -Remicade ®, infliximab's biosimilar- Inflectra®, Remsima®, or any other biosimilar or branded biological agent All anti TNF alpha agents will have to be prescribed in the same administration modality and dosing regimen than in the control group and according to the Summary of Product Characteritics (SmPC) MTX: 15 mg a week orally: on a fixed day of the week defined for each patient In patients receiving an anti TNF alpha according to the SmPC, MTX will be initiated within 7 days after the start of the anti TNF alpha agent
  Interventions: Drug: Methotrexate
- Control group (Placebo Comparator): Use of placebo- MTX in psoriasis patients receiving anti TNF alpha agent according to the approved indication: etanercept- Enbrel®, adalimumab- Humira ®, infliximab -Remicade ®, infliximab's biosimilar- Inflectra®, Remsima®, or any other biosimilar or branded biological agent
  All anti TNF alpha agents will have to be prescribed in the same administration modality and dosing regimen than in the experimental group and according to the SmPC Placebo-MTX orally: on a fixed day of the week defined for each patient In patients receiving an anti TNF alpha according to the SmPC, MTX-placebo will be initiated within 7 days after the start of the anti TNF alpha agent
  Interventions: Drug: Methotrexate Placebo

INTERVENTIONS:
Drug: Methotrexate — Use of low dose methotrexate (MTX) in psoriasis patients receiving an anti TNF alpha agent
  Arms: Experimental group
Drug: Methotrexate Placebo — Use of placebo- MTX in psoriasis patients receiving anti TNF alpha agent according to the approved indication
  Arms: Control group

SUMMARY:
The overall purpose of this trial is to assess efficacy and safety of the combination of low doses of Methotrexate (MTX) with anti Tumor Necrosis Factor (TNF) alpha to improve initial efficacy and maintenance rate of anti-TNF alpha treatment in patients with psoriasis.

DETAILED DESCRIPTION:
The combination of an anti-TNF alpha and methotrexate may also prevent the development of antibodies to anti TNF alpha. Observational studies indicated that MTX dose-dependently inhibits the development of anti-drug antibodies and could reduce the accelerated clearance of biological agents associated with loss of therapeutic response in inflammatory diseases. Reduced ADA development influence positively clinical response and therefore likely drug maintenance through optimizations of drug pharmacokinetics and serum anti TNF alpha trough concentrations.

In psoriasis, there is no prospective evaluation of the combination MTX-anti TNF alpha to help to maintain long-term efficacy for all anti TNF alpha. Long-term maintenance treatment with the combination of MTX and infliximab was reported in one small retrospective cohort study of psoriasis patients experiencing a loss of response to infliximab (55). In total 23 patients received as a rescue either azathioprine (5 patients) or weekly MTX (18 patients) (7.5 to 15 mg, average 11.66 mg) in combination with infliximab. After a mean follow up of 26.5 months, only 2 patients on MTX combination stopped infliximab for loss of response which is lower compared to the 50% loss of response observed with infliximab monotherapy (55).

The combination of anti TNF alpha and MTX was also retrospectively assessed in observational studies. Most of them suggest that the systematic combination of MTX to biologic since the anti TNF alpha initiation improve survival rate of biologics (21, 24, 29, 30, 31). A retrospective cohort study including 93 patients treated with infliximab for psoriasis showed that concomitant MTX at an average weekly dose of dose of 7.5 to 17.5 mg of MTX enhanced the maintenance of response and prolonged drug survival (by a mean ± SD of 19.5 ± 8.1 months, P = 0.034) (23). In addition, time until first infliximab dose escalation was delayed in patients receiving MTX (by a mean ± SD of 12.0 ± 6.1 months, P =0 .037). In the same study, after 2 years of treatment, 25% of patients without MTX were still under the initial infliximab regimen versus 40% of patients receiving a combination of infliximab with MTX (30).

The ability of MTX to prolong drug survival was also suggested in psoriatic arthritis in several observational studies (26, 27, 52, 56). In a longitudinal observational study, the 1-year retention rate of anti-tumor necrosis factor alpha medications in patients with RA and PsA were 65.4% and 77.3%, respectively with concomitant MTX associated with a better drug survival (52). In this study, the combination with MTX was also associated with a crude 1-year survival of 85% in PsA versus 70% without concomitant MTX, p=0.02 (52). In the Danish biologics registry DANBIO, male sex, CRP level >10 mg/liter, concomitant methotrexate use, and low patient health visual analog scale score at baseline were associated with longer drug survival in PsA patients (27).

To summarize, there is a need to improve drug survival as well as level of response rates with biologics, especially for psoriasis patients. Low doses methotrexate when combining to biologics could be an option in psoriasis patients to solve such crucial issues.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* Patients with moderate to severe chronic plaque psoriasis with or without psoriatic arthritis AND who had started any first line of anti TNF alpha according to the labeling of these drugs BEFORE the study (i. e. the study will be restricted to anti TNF alpha naïve patients (first course). Patients who have been previously treated with any other non anti TNFA alpha biopharmaceutical (ustekinumab or anti IL17- secukinumab, ixekizumab, brodalumab) as a first line of biotherapy for psoriasis could be enrolled) after a wash out period of at least 5 half life time of the drug i.e. 16 weeks before inclusion
* No significant anomalies from a blood sampling performed within 15 days before patient selection that could lead to MTX contraindication
* Patients with an EARLY start of anti TNF alpha, i. e. within the 7 days preceding the first study drug (methotrexate or placebo) administration
* Male or female patients agreeing to use a reliable method of birth control during the study

  * Male patients agreeing to use a reliable method of birth control during the study i. e. preservative and for at least 6 months following the last dose of investigational product, the patient's partner treated by methotrexate must be notified of the teratogenic risk of methotrexate and should be under effective contraception throughout the study
  * Female patients:

Are women of childbearing potential who are negatively tested for pregnancy and agree to use a reliable method of birth control (every month) or remain abstinent during the study and for at least 6 months following the last dose of investigational product, whichever is longer. Methods of contraception considered acceptable include oral contraceptives, contraceptive patch, intrauterine device, vaginal ring.

And Negative serum b-Human Chorionic Gonadotrophin (B-HCG) test at screening Or

Women of non-childbearing potential, defined as:

Women who have had a surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) Or Women > = 60 years of age Or Women >=40 and < 60 years who have had a cessation of menses for >=12 months and a follicule stimulating hormone (FSH) test confirming non - childbearing potential

* Patients with previous failure or intolerance but no absolute contraindication to previous methotrexate medication for psoriasis can be enrolled, on the condition that methotrexate (whatever the dose) has been stopped at least two months before the inclusion.
* For patients who have never been previously treated with MTX, taking a test dose of MTX (2.5 mg to 5 mg) with normality of the laboratory tests conducted one week to remove a reaction idiosynchrasie before inclusion in the protocol
* Patients should be affiliated to the French Social Security system
* Patients who have given written consent for the study

Exclusion Criteria:

* Patients with isolated pustular, erythrodermic and or guttate forms of psoriasis
* Patients with prior use of any anti TNF alpha
* Patients who have known active liver disease (with the exception of a simple liver steatosis, transaminases and/or alkaline phosphatases > 2 ULM ) or history of liver disease in the past 2 years, whatever the related diagnosis but which could interfere with MTX safety and according to the summary of the SmPC
* Intake of restricted medications (cf section VIII.5.) or other drugs considered likely to interfere with the safe conduct of the study, as assessed by the investigator and according to the Summary of the Product Characteristics (SmPC), including any drug intakes that could interfere with methotrexate metabolism or that could enhance liver and /or hematologic toxicity and according to the SmPC
* Patient with evidence or positive test for HIV, Hepatitis C virus, Hepatitis B virus (patients who are negative for hepatitis B surface antigen but positive for anti-hepatitis B anti body (HBsAb+ and HBcAb+) and negative for serum HBV DNA may participate in the study
* High alcohol intake defined as more than 60 g of daily intake (approx daily intake of 0.5 l of wine or equivalent),
* Patients who have a known allergy or hypersensitivity to MTX
* Patients who have a known serious adverse event to MTX prior to the trial leading to MTX discontinuation in the past
* Presence of significant hematologic or renal disorder or abnormal laboratory values at screening that, in the opinion of the investigator is associated with an unacceptable risk to the patient to participate in the study
* Clinical laboratory test results at screening that are outside a normal reference rating for the population and are considered clinically significant, or/and have any of the following specific abnormalities:

  * Total white blood cell count <3G/L
  * Neutrophil count < 1.5 G/l
  * Lymphocytes count < 0.5G/l
  * . Platelet count < 100 G/l
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>3 times the upper limit of normal (ULM)
  * Hemoglobin <8.5g/dL (85.0 g/L)
  * Creatinine clearance <40ml/min (Cockcroft formula)
* For women: pregnant or breast feeding
* Patients who have an active or serious infection or history of infections (bacterial, viral, fungal or mycobacteria), requiring hospitalization or intra venous anti-infectives infusion within 4 weeks prior to the baseline,
* Patients who have primary or secondary active immunodeficiency
* Patients who had live vaccine administration within 4 weeks prior to baseline
* Patients who have any current or active cancer (with the exception of patient with successfully treated basal cell carcinoma or in situ cervix carcinoma)
* Patients who had history of malignancy within 5 years prior to the trial that could contraindicate the use of an immunosuppressant
* Patients who will not be available for protocol which require study visits or procedures
* Patients who is not affiliated to the French Social Security system
* Patients unable to give informed consent and/or comply with all required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Loss of response from the index anti TNF alpha | 24 months
  The primary endpoint is the loss of response from the index anti TNF alpha is defined as the time (or time interval) between baseline and the loss of PASI 75 response (loss of the improvement of at least 75% of the initial disease severity (loss of PASI 75).The respective loss of response between MTX and placebo in combination with the anti TNF alpha will be assessed for both groups during month (M) 24.
  The survival curves will be compared between the groups (MTX and placebo) using the log rank test.

SECONDARY OUTCOMES:
Initial response to the index anti TNF alpha | 4 months
  measured by the PASI score assessed at M3 (etanercept) or M4 (others anti-TNF alpha).
  It will be categorized as follows:
  * Efficacy: achievement of at least 75% improvement from baseline PASI score i. e. PASI >= 75 at M3 (etanercept) or M4 (others anti-TNF alpha).
  * Intermediate response: achievement of a PASI response between 50% and 75% improvement from baseline PASI score at M3 (etanercept) or M4 (others anti-TNF alpha).
  * Treatment failure: less than 50% improvement from baseline PASI score i. e. PASI < 50 at M3(etanercept) or M4 (others anti-TNF alpha).
  The initial response rates will be assessed in the whole population and also separately for each anti TNF alpha agent at M3 (etanercept) or M4 (others anti-TNF alpha).
The maintenance of response rates proportion of patients who are still treated with the index anti TNF alpha agent without any drug adjustment | 24 months
  It will be assessed after M3 (etanercept) or M4 (others anti-TNF alpha) according to:
  The maintenance of response rates will be assessed in the whole population and also separately for each anti TNF alpha agent at M6, M9, M12, M18, M24.physiological parameter,
Assessment of patient's quality of life using the Dermatology Quality of Life (DLQI) | 24 months
  DLQI is a dermatology-specific Quality of Life instrument . Assessment will be performed at baseline, M3 (etanercept) or M4 (others anti-TNF alpha), M9, M12, M18, M24.
  - Treatment satisfaction assessment for medication will be assessed at M3 (etanercept) or M4 (others anti-TNF alpha), M9, M12, M18, M24.
Assessment of the study drugs 'safety: number of Adverse Events (AE) and serious adverse events (SAE), as well as the proportion of discontinuation due to AEs and/or SAEs | 24 months
Assessment of the sutdy drugs' (MTX and MTX placebo) tolerability by measuring the possible changes in vital signs and occurence of AE such as asthenia, digestive tolerance, headache. | 24 months
  Vital signs, temperature and clinical examination will be assessed at M3 (etanercept) or M4 (others anti-TNF alpha), M9, M12, M18, M24 . Changes with blood safety laboratory analysis (hematology, liver and renal tests recommended by SmPC and pregnancy tests) will also be assessed at M1, M2, M3 (etanercept) or M4 (others anti-TNF alpha), M6, M9, M12, M15, M18, M21, M24

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided